CLINICAL TRIAL: NCT06363214
Title: Impact of Patient Blood Management (PBM) at the Schulthess Clinic A Quality Assurance and Quality Control Project in Major Orthopaedic and Spine Surgery
Brief Title: Impact of Patient Blood Management (PBM) at the Schulthess Clinic
Acronym: PBM
Status: Not yet recruiting | Type: Observational
Sponsor: Schulthess Klinik (Other)
Responsible Party: Principal Investigator, Christoph Hofer, Head of Anesthesia, Professor, Principal Investigator, Schulthess Klinik
Other Study IDs: ANEST-0002
Record Dates: First submitted 2024-04-09; First posted 2024-04-12 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Patient Blood Management
Keywords: blood transfusion; orthopedic surgery; coagulation
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Patient blood management — Perioperative optimization of hemoglobin level, perioperative minimization of blood loss, increase of anemia tolerance

SUMMARY:
Aim of this study is to analyze the transfusion requirements of allogenic blood products at the Schulthess Clinic for patients that had major orthopedic or major spine surgery between 2019 and 2024 order to identify patients at risk for transfusion. Moreover, impact of transfusion requirements and other measures of PBM on patient outcomes will be assessed. These data are required to further improve PBM at the Schulthess Clinic.

DETAILED DESCRIPTION:
At the Schulthess Clinic a significant reduction of RBC's, fresh frozen plasma (FFP) and platelets transfusion could be observed between 2018 and 2022 during the stepwise introduction of PBM for all patients undergoing major orthopedic and spine surgery. RBC, FFP and PT transfusion declined by 76.3%, 73.5% and 99.2% over the 5-year period. Unfortunately however, at the moment no detailed analysis with respect to risk factors for transfusion, specific interventions or outcomes is available. The hypothesis is that the already known reduction of allogenic blood product transfusion at the Schulthess Clinic can be attributed to patients undergoing major primary joint arthroplasties, revision operations and major spine surgery. We assume that patient and procedure related risk factors over time did not significantly change while we expect a major impact of changed transfusion requirements and the stepwise PBM implementation on patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing primary joint arthroplasties or revision surgery: CHOP Code: 81.51, 81.52, 81.52, 81.54
* Patients undergoing major spine surgery: CHOP Code: 7A.6, 7A.7

Exclusion Criteria:

* Patients who did not sign general informed consent

Ages: 16 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing elective major orthopedic or spine surgery at the Schulthess Clinic between 2019 and 2024.
Sampling Method: Non-Probability Sample
Enrollment: 16000 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Perioperative transfusion rates | 2019-2024
  Administration of red blood cells, fresh frozen plasma and platelet concentrates (units)
Risk factors for perioperative transfusion Risk factors for perioperative transfusion Risk factorsfor perioperative transfusion | 2019-2024
  Identification of patient groups with increased transfusion rates

SECONDARY OUTCOMES:
Perioperative rates of coagulation products administered | 2019-2024
  Administration of prothrombin complex, fibrinogen, other coagulation factors
Clinical outcomes | 2019-2024
  * Infections: Wound, sepsis, drug-resistant, Clostridium difficilis.
  * Ischemic events: TIA, cerebrovascular, myocardial
  * Thrombotic: Deep venous thrombosis (DVT), pulmonary embolism (Barrie et al.)
  * Renal failure
  * Pulmonary failure

CONTACTS AND LOCATIONS:
Overall Officials: Christoph K Hofer, MD, Principal Investigator — Schulthess Klinik

IPD SHARING:
Plan to Share IPD: No